CLINICAL TRIAL: NCT01716702
Title: A Feasibility Study of an Online Intervention for Sexual Rehabilitation in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDHA-RS/2013-076
Record Dates: First submitted 2012-10-16; First posted 2012-10-30 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Psychosocial Intervention; Sexual Rehabilitation; Online Intervention
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Couples Prostate Cancer Support Group (Experimental): The participants in the support group will receive 6 weekly online intervention sessions with a professional facilitator. In addition participants will be asked to complete relationship-enhancement exercises and readings in between sessions.
  Participants will be asked to complete questionnaires at three time points: 1)pre-intervention (baseline) 2) post-intervention (7 weeks), and 3) post intervention (13 weeks).
  Interventions: Behavioral: Couples Prostate Cancer Support Group
- Wait-List Control (No Intervention): Participants will be asked to complete questionnaires at three time points: 1)week 1 2) week 7, and 3) week 13.

INTERVENTIONS:
Behavioral: Couples Prostate Cancer Support Group — The participants in the experimental group will receive 6 weekly online intervention sessions with a professional facilitator. In addition participants will be asked to complete relationship-enhancement exercises and readings in between sessions.
  In the experimental group, participants will be asked to complete questionnaires at three time points: 1)pre-intervention (baseline) 2) post-intervention (7 weeks), and 3) post intervention (13 weeks).
  In the waitlist group, participants will not participate in the support group. Participants will be asked to complete questionnaires at three time points: 1)pre-intervention (baseline) 2) post-intervention (7 weeks), and 3) post intervention (13 weeks).
  Arms: Couples Prostate Cancer Support Group

SUMMARY:
Background: Prostate cancer (PCa) is the most common cancer for men. When treated early enough it is typically curable. However, common treatments, such as radical prostatectomy and radiation therapy, often result in significant negative outcomes with regard to sexual, psychological and social function. Both men and partners have identified the need for more information and support to address sexual health concerns after treatment. However, very few sexual rehabilitation interventions have been developed and rigorously assessed.

Purpose: The investigators propose to develop and pilot test a new program to meet the sexual health needs of men with PCa and their partners using an online, professionally facilitated education/support program. The goals of the program are to improve sexual function, intimacy and mood for men and their partners after treatment for localized PCa. The program will be offered through Cancer Chat Canada, an existing and well-tested Canadian platform for professionally facilitated support group programs.

What Participants Can Expect: A total of 24 men and their female partners (48 individuals) will be recruited and assigned to one of two groups. The first group will participate in the program immediately; the second group will be offered the program after a 5-month delay. The decision about which group will start immediately and which later will be made randomly (by chance). Both groups of men and partners will be asked to complete questionnaires three times and, at the end of the program, to provide the researchers feedback about how satisfied they were with the program, the changes they made, things they learned as a result of the program, and suggestions for improving the program. Participants must have access to a computer, an Internet connection and be willing to attend online, chat room meetings each week for 1.5 hours for 6 weeks.

Implications: Sexual rehabilitation is a high need for men affected by PCa, but is difficult to access. The investigators hope to improve access to sexual health care through this study.

ELIGIBILITY:
Inclusion Criteria:

* Men who have been treated for localized prostate cancer
* AND men must be 6-36 months post-prostatectomy or radiation (as primary treatment) of prostate cancer
* Must have a heterosexual, co-cohabiting partner who is willing to participate
* Must speak and read English
* Must be able to use a computer and have internet access

Exclusion Criteria:

* Homosexual couples will not be included in this study
* Major self-reported psychiatric illness
* Couples who screen below 30 on the DAS (Dyadic Adjustment Scale)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Function from Baseline to 13 weeks | Pre-Intervention (Week 1); Post-Intervention (Week 7); 3 Months Post-Intervention (Week 13)

SECONDARY OUTCOMES:
Change in Personal Assessment of Intimacy and Relationships from baseline to 13 weeks | Pre-Intervention (Week 1); Post-Intervention (Week 7); 3 Months Post-Intervention (Week 13)

OTHER OUTCOMES:
Change in Profile of Mood States Short Form from baseline to 13 weeks | Pre-Intervention (Week 1); Post-Intervention (Week 7); 3 Months Post-Intervention (Week 13)
  This tool assesses psychological distress across 6 domains: fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L McLeod, R.N., Ph.D., Principal Investigator — Capital District Health Authority & Dalhousie University; Richard J Wassersug, Ph.D., Principal Investigator — University of British Columbia; Karen Fergus, Ph.D., C. Psych., Principal Investigator — Sunnybrook Odette Cancer Centre & York University; John Robinson, Ph.D., C. Psych., Principal Investigator — Tom Baker Cancer Centre & University of Calgary; John Oliffe, R.N, Ph.D., Principal Investigator — University of British Columbia
Locations (1):
- Capital District, Halifax, Nova Scotia, Canada